CLINICAL TRIAL: NCT07210138
Title: The Clinical Investigation of PerioGard (Test) Regimen Compared to Control Regimen in Reducing Plaque and Gingivitis - a Three-month Study in Thailand
Brief Title: Clinical Investigation of PerioGard (Test) Regimen
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRO-2025-05-GUM-RGM-THA-YPZ
Record Dates: First submitted 2025-09-29; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-06

CONDITIONS: Gingivitis
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Test regimen (Experimental): Test Regimen: toothpaste, mouthwash and toothbrush
  Interventions: Drug: PeriGuard regimen
- Control regimen (Active Comparator): Control regimen: toothpaste, mouthwash and toothbrush
  Interventions: Drug: Colgate Dental Cream regimen

INTERVENTIONS:
Drug: PeriGuard regimen — 0.45% Stannous Fluoride Toothpaste, CPC-Zinc Fluoride Mouthwash, Gummy Toothbrush
  Arms: Test regimen
Drug: Colgate Dental Cream regimen — Colgate Cavity Protection Toothpaste, Fluoride Mouthwash,Colgate Extra Clean Soft-Bristled Toothbrush
  Arms: Control regimen

SUMMARY:
The objective of this three-month clinical research study is to evaluate the clinical efficacy of the PerioGard (test) regimen (0.45% SnF-HW Toothpaste, CPC-Zinc-Fluoride Mouthwash, Gummy Toothbrush) compared to the control regimen (regular fluoride toothpaste, fluoride mouthwash, flat-trim toothbrush) in reducing gingivitis and dental plaque in adults

ELIGIBILITY:
Inclusion Criteria:

* Subjects, ages 18-70, inclusive.
* Availability for the three-month duration of the clinical research study.
* Good general health.
* Minimum of 20 uncrowned permanent natural teeth (excluding third molars).
* Initial gingivitis index of at least 1.0 as determined by the use of the Loe and Silness Gingival Index.
* Initial plaque index of at least 1.5 as determined by the use of the Quigley and Hein Plaque Index (Turesky Modification).
* Signed Informed Consent Form.

Exclusion Criteria:

* Presence of orthodontic bands.
* Presence of partial removable dentures.
* Tumor(s) of the soft or hard tissues of the oral cavity.
* Advanced periodontal disease (purulent exudate, tooth mobility, and/or extensive loss of periodontal attachment or alveolar bone).
* Five or more carious lesions requiring immediate restorative treatment.
* Antibiotic use any time during the one-month period prior to entry into the study.
* Participation in any other clinical study or test panel within the one month prior to entry into the study.
* Dental prophylaxis during the past two weeks prior to baseline examinations.
* History of allergies to oral care/personal care consumer products or their ingredients.
* On any prescription medicines that might interfere with the study outcome.
* An existing medical condition that prohibits eating or drinking for periods up to 4 hours.
* History of alcohol or drug abuse.
* Pregnant or lactating subjects.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2025-08-18 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Measurement of Loe-Silness Gingival Index score | baseline, 1 week, 4 week and 3 month
  Loe-Silness Gingival Index score from 0 to 3 will be assigned by the examining dentist to all scoreable surfaces of the maxillary and mandibular teeth using a dental light and dental mirror. A whole mouth mean score for each subject will be determined by adding the values given by the examining dentist to each scoreable surface and dividing that number by the total number of surfaces scored.
Measurement of Quigley-Hein Plaque Index score | baseline, 1 week, 4 week and 3 month
  First using a red dye solution to disclose the plaque, a Quigley-Hein Plaque Index score of 0 to 5 will be assigned to all scoreable disclosed surfaces of the maxillary and mandibular teeth using a dental light and dental mirror. A whole mouth score for each subject will be determined by adding the values given by the dental examiner to each scoreable surface and dividing that number by the total number of surfaces scored.

CONTACTS AND LOCATIONS:
Overall Officials: Terdphong Triratana, DDS, Principal Investigator — Mahidol University
Locations (1):
- Mahidol University, Ratchathewi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No